CLINICAL TRIAL: NCT01732913
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Idelalisib (GS-1101) in Combination With Rituximab for Previously Treated Indolent Non-Hodgkin Lymphomas
Brief Title: Efficacy and Safety of Idelalisib (GS-1101) in Combination With Rituximab for Previously Treated Indolent Non-Hodgkin Lymphomas
Acronym: Yosemite
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-313-0124
Record Dates: First submitted 2012-11-14; First posted 2012-11-26 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2017-03

CONDITIONS: Indolent Non-Hodgkin's Lymphomas
Keywords: iNHL; indolent NHL; follicular lymphoma; CAL-101; Rituximab; Small lymphocytic lymphoma; lymphoplasmacytoid lymphoma; Waldenstrom macroglobulinemia; LPL; WM; Marginal zone lymphoma; MZL; SLL; FL; GS-1101; idelalisib
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; idelalisib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rituximab + idelalisib (Experimental): Participants will receive rituximab + idelalisib.
  Interventions: Drug: Rituximab; Drug: Idelalisib
- Rituximab + Placebo (Placebo Comparator): Participants will receive rituximab + placebo. Following confirmation of iNHL disease progression by the independent review committee and unblinding, participants may be eligible to receive open-label idelalisib 150 mg twice daily.
  Interventions: Drug: Placebo; Drug: Rituximab; Drug: Idelalisib

INTERVENTIONS:
Drug: Placebo — Tablets administered orally twice daily
  Arms: Rituximab + Placebo
Drug: Rituximab — 375 mg/m^2 administered intravenously weekly for 4 weeks, then every 8 weeks (up to a total of 8 infusions)
  Other Names: Rituxan®; MabThera®
Drug: Idelalisib — 150 mg tablets administered orally twice daily
  Other Names: GS-1101; CAL-101; Zydelig®

SUMMARY:
The primary objective of this study is to evaluate the effect of the addition of idelalisib to rituximab on progression-free survival (PFS) in adults with previously treated indolent non-Hodgkin lymphoma (iNHL).

An increased rate of deaths and serious adverse events (SAEs) among participants with front-line chronic lymphocytic leukemia (CLL) and early-line iNHL treated with idelalisib in combination with standard therapies was observed by the independent data monitoring committee (DMC) during regular review of 3 Gilead Phase 3 studies. Gilead reviewed the unblinded data and terminated this study in agreement with the DMC recommendation and in consultation with the US Food and Drug Administration (FDA).

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of B-cell iNHL, with histological subtype limited to the following:

  1. Follicular lymphoma (FL) Grade 1, 2, or 3a
  2. Small lymphocytic lymphoma (SLL) with absolute lymphocyte count < 5 x 10^9/L at the time of diagnosis
  3. Lymphoplasmacytoid lymphoma/Waldenström macroglobulinemia (LPL/WM)
  4. Marginal zone lymphoma (MZL) (splenic, nodal, or extra-nodal)

Key Exclusion Criteria:

* History of lymphoid malignancy other than those allowed per inclusion criteria
* Ongoing drug-induced liver injury, active hepatitis C, active hepatitis B , alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension.
* Received previous treatment with rituximab that was not effective.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2013-01-16 (Actual); Primary Completion 2016-05-18 (Actual); Study Completion 2016-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (103):
- United States (32):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - City of Hope Cancer Center, Duarte, California
  - Saint Jude Heritage Healthcare, Fullerton, California
  - Pacific Shores Medical Group, Long Beach, California
  - UCLA Medical Center, Los Angeles, California
  - Cancer Care Associates, Redondo Beach, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Central Coast Medical Oncology Group, Santa Maria, California
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists and Research Institute, Fort Myers, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Cancer Center of Kansas, Wichita, Kansas
  - Wayne State University, Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - MetroHealth Medical Center, Cleveland, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Prairie Lakes Healthcare System, Watertown, South Dakota
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Texas Oncology, P.A., Bedford, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Center for Cancer and Blood Disorders, PC, Fort Worth, Texas
  - Shenandoah Oncology Associates, PC, Winchester, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - Haematology and Oncology Clinics of Australia at Chermside, Milton, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Saint Vincent's Hospital, Fitzroy, Victoria
  - Western Hospital, Footscray, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Adelaide Cancer Centre, Kurralta Park
  - Fiona Stanley Hospital, Murdoch
- Fakultní nemocnice Hradec Králové, Hradec Králové, Czechia
- France (10):
  - University Hospital of Bordeaux, Pessac, Aquitaine
  - Centre Hospitalier Régional Universitaire de Lille, Hôpital Claude Huriez, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire Brest, Brest
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Centre Hospitalier de Versailles, Le Chesnay
  - Centre Léon Bérard, Lyon
  - Hôpital Hôtel-Dieu, Nantes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers Hôpital de la Milétrie, Poitiers
  - Hôpital Necker-Enfants Malades, Paris, Île-de-France Region
- Germany (2):
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen, Baden-Wurttemberg
  - Gemeinschaftspraxis Dres. Söling Und Siehl, Kassel, Hesse
- Hungary (5):
  - Debreceni Egyetem Orvos-és Egészségtudományi Centrum, Debrecen, Hajdú-Bihar
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County
  - Markusovszky Egyetemi Oktatókórház, Szombathely, Vas County
  - Semmelweis Egyetem, Budapest
  - Országos Onkológiai Intézet, Budapest
- Israel (2):
  - Hadassah Medical Organization, Ein Kerem, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Italy (5):
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico S.Orsola-Malpighi, Bologna
  - Azienda Ospedaliero Universitaria (AOU) "Maggiore della Carita" di Novara, Novara
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro
  - Centro di Riferimento Oncologico di Aviano, Pordenone
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Japan (13):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Kyushu Cancer Center, Minamiku, Fukuoka
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - National Hospital Organization Kumamoto Medical Center, Chuo-ku, Kumamoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka City University Hospital, Osaka, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Toranomon Hospital, Minato-ku, Tokyo
- Poland (3):
  - Malopolskie Centrum Medyczne S.C., Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Ministerstwa Spraw Wewnetrznych z Warminsko-Mazurskim, Olsztyn
  - Centrum Onkologii i Hipertermii, Warsaw
- Hospital Geral de Santo António do Centro Hospitalar do Porto, Porto, Portugal
- Institutul Clinic Fundeni, Bucharest, Romania
- Russia (6):
  - Nizhny Novgorod Regional Clinical Hospital n.a. N.A. Semashko, Nizhny Novgorod
  - Ryazan Regional Clinical Hospital, Ryazan
  - Saint Petersburg I.P. Pavlov State Medical University, Saint Petersburg
  - FSI "V.A. Almazov Federal Centre of Heart, Blood and Endocrinology of Rosmedtechnologies", Saint Petersburg
  - Saratov State Medical University, Saratov
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- Singapore (3):
  - Singapore General Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
  - Gleneagles Medical Centre, Singapore
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (2):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitari Germans Trias i Pujol, Badalona
- Skånes Universitetssjukhus, Malmö, Malmo, Sweden
- Taiwan (2):
  - Chang Gung Memorial Hospital (CGMH), Kaohsiung City
  - Tri-Service General Hospital, Taipei
- United Kingdom (3):
  - Barts and The London NHS Trust, London, England
  - Mount Vernon Hospital, Middlesex
  - Sunderland Royal Infirmary, Sunderland

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the North America, Europe, and Asia Pacific. The first participant was screened on 16 January 2013. The last study visit occurred on 18 May 2016.
Pre-assignment Details: 385 participants were screened.
Groups:
- Idelalisib + Rituximab: Idelalisib (Zydelig®) 150 mg tablet orally twice daily + rituximab 375 mg/m^2 intravenously starting on Day 1 for a total of 8 infusions
- Placebo + Rituximab: Placebo tablet orally twice daily + rituximab 375 mg/m^2 intravenously starting on Day 1 for a total of 8 infusions
Period: Overall Study
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Started | 198 | 97
Completed (Completed = reached primary efficacy endpoint of progressive disease or death) | 42 | 28
Not Completed | 156 | 69
Not completed — Study Terminated by Sponsor | 105 | 55
Not completed — Withdrawal by Subject | 27 | 4
Not completed — Physician Decision | 14 | 7
Not completed — Other | 7 | 1
Not completed — Initiation of Other Anti-Cancer Therapy | 3 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Analysis Set: all participants who were randomized regardless of whether they received any study treatment
Groups:
- Idelalisib + Rituximab: Idelalisib 150 mg tablet orally twice daily + rituximab 375 mg/m^2 intravenously starting on Day 1 for a total of 8 infusions
- Total: Total of all reporting groups
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab | Total
Number analyzed (Participants) | 198 | 97 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11.4) | 67 (11.4) | 65 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 48 | 147
  Male | 99 | 49 | 148
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 35 | 17 | 52
  Black or African American | 5 | 4 | 9
  White | 123 | 54 | 177
  Other | 3 | 3 | 6
  Not Permitted | 32 | 19 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 3 | 15
  Not Hispanic or Latino | 150 | 75 | 225
  Unknown or Not Reported | 36 | 19 | 55
Region of Enrollment [Count of Participants; unit: Participants]
  Russian Federation | 7 | 2 | 9
  Singapore | 5 | 4 | 9
  Romania | 1 | 0 | 1
  Hungary | 24 | 6 | 30
  United States | 65 | 34 | 99
  Japan | 23 | 9 | 32
  United Kingdom | 3 | 1 | 4
  Portugal | 3 | 1 | 4
  Spain | 6 | 0 | 6
  Czech Republic | 2 | 0 | 2
  Sweden | 6 | 2 | 8
  Taiwan | 1 | 1 | 2
  Poland | 5 | 7 | 12
  Korea, Republic of | 4 | 2 | 6
  Italy | 7 | 4 | 11
  Israel | 3 | 0 | 3
  Australia | 7 | 6 | 13
  France | 25 | 17 | 42
  Germany | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is defined as the interval from randomization to the earlier of the first documentation of definitive indolent non-Hodgkin lymphoma (iNHL) disease progression or death from any cause. PFS was to be assessed by an independent review committee (IRC).
Population: Due to the early termination of the study, efficacy data were not available for all participants, and therefore the prespecified analyses were not conducted.
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Response Rate
Description: Overall Response Rate (ORR) is defined as the proportion of participants who achieve a complete response or partial response (or very good partial response or minor response for participants with Waldenstrom's). ORR was to be assessed by an IRC.
Population: as for outcome 1
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Lymph Node Response Rate
Description: Lymph node response rate is defined as the proportion of participants who achieve ≥ 50% decrease from baseline in the sum of the products of the greatest perpendicular diameters of index lesions. Lymph node response rate was to be assessed by an IRC.
Population: as for outcome 1
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Complete Response Rate
Description: Complete response rate is defined as the proportion of participants who achieve a complete response. Complete response rate was to be assessed by an IRC.
Population: as for outcome 1
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the interval from randomization to death from any cause.
Population: Due to the early termination of the study, efficacy data were not mature for all participants, and therefore the prespecified analyses were not conducted.
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 27 months plus 30 days
Description: Safety Analysis Set
Arm/Group | Idelalisib + Rituximab | Placebo + Rituximab
Serious Adverse Events (participants affected / at risk) | 103/198 | 11/95
Other Adverse Events (participants affected / at risk) | 189/198 | 83/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Rituximab (N=198) | Placebo + Rituximab (N=95)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 2
Pericarditis (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 8 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 18 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Salivary gland disorder (Gastrointestinal disorders) | 0 | 1
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 2 | 0
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Gait disturbance (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 9 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 3 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0
Jaundice (Hepatobiliary disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 2 | 0
Eczema herpeticum (Infections and infestations) | 1 | 0
Fungaemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster meningomyelitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 19 | 0
Sepsis (Infections and infestations) | 5 | 0
Septic shock (Infections and infestations) | 1 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 4 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 11 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 3 | 0
Transient ischaemic attack (Nervous system disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Rituximab (N=198) | Placebo + Rituximab (N=95)
Anaemia (Blood and lymphatic system disorders) | 12 | 6
Neutropenia (Blood and lymphatic system disorders) | 25 | 5
Abdominal pain (Gastrointestinal disorders) | 20 | 4
Constipation (Gastrointestinal disorders) | 28 | 13
Diarrhoea (Gastrointestinal disorders) | 88 | 18
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 3
Nausea (Gastrointestinal disorders) | 50 | 12
Vomiting (Gastrointestinal disorders) | 29 | 7
Asthenia (General disorders) | 15 | 9
Chills (General disorders) | 11 | 4
Fatigue (General disorders) | 41 | 20
Oedema peripheral (General disorders) | 14 | 5
Pyrexia (General disorders) | 50 | 11
Bronchitis (Infections and infestations) | 9 | 6
Nasopharyngitis (Infections and infestations) | 10 | 6
Upper respiratory tract infection (Infections and infestations) | 23 | 8
Urinary tract infection (Infections and infestations) | 13 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 36 | 20
Alanine aminotransferase increased (Investigations) | 65 | 0
Aspartate aminotransferase increased (Investigations) | 56 | 0
Gamma-glutamyltransferase increased (Investigations) | 11 | 1
Transaminases increased (Investigations) | 12 | 1
Weight decreased (Investigations) | 20 | 1
Decreased appetite (Metabolism and nutrition disorders) | 26 | 2
Dehydration (Metabolism and nutrition disorders) | 11 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 3
Dizziness (Nervous system disorders) | 12 | 6
Headache (Nervous system disorders) | 30 | 12
Anxiety (Psychiatric disorders) | 10 | 3
Insomnia (Psychiatric disorders) | 21 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 25 | 4
Rash (Skin and subcutaneous tissue disorders) | 38 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16 | 2
Hypertension (Vascular disorders) | 12 | 2

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, efficacy data were not available for all participants, and therefore the prespecified analyses were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years